CLINICAL TRIAL: NCT02022059
Title: Prospective Monocentric Study on the Efficacy of Lidocain Spray for Patient Comfort During Nasogastric Tube Insertion in Enteral Nutrition: the Xylonut Trial
Brief Title: Prospective Monocentric Study on the Efficacy of Lidocain Spray for Patient Comfort During Nasogastric Tube Insertion in Enteral Nutrition
Acronym: Xylonut
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-AOI-12
Record Dates: First submitted 2013-12-06; First posted 2013-12-27 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): patient nécessitant une SNG pour nutrition entérale bénéficiant d'une pré-médication par vaporisateur de lidocaïne lors de l'insertion (group A = lidcoaine)
  Interventions: Drug: Lidocaine = group A
- Placebo (Placebo Comparator): Patient requiring a SNG for nutrition entérale benefiting from a pre-medication by placebo during the insertion (group B)
  Interventions: Drug: Group B placebo

INTERVENTIONS:
Drug: Lidocaine = group A — Patient requiring a SNG for nutrition entérale benefiting from a pre-medication by spray of lidocaïne during the insertion (group A = lidocaine)
  Arms: Lidocaine
Drug: Group B placebo — Patient requiring a SNG for nutrition entérale benefiting from a pre-medication by placebo during the insertion
  Arms: Placebo

SUMMARY:
Enteral nutrition is the treatment of choice for malnourish patient. Nasogastric tube (NGT) is although a common act. Unfortunately, this procedure can be painful. Also, many patients will need many NGT re-insertion. Therefore, the investigators need to increase the acceptability of this procedure by increasing comfort during NGT passage. Professionals guidelines of HAS (recommendations professionnelles de bonne pratiques de soins) and SFNEP (Société Française de Nutrition Clinique et Métabolisme) talk about the possibility of using local anesthesic without ordering their use. However, NGT tube insertion is often put without pre-medication in the face of an accumulating body of evidence indicating that local anesthetic prior NGT insertion decrease discomfort of the procedure. On the other hand, these studies have been done in the emergency room with NGT of a bigger gauge and for many reasons except enteral nutrition.

The investigators primary objective of this prospective monocentric study is to evaluate the efficacy (patient comfort) of lidocaine 5 % spray versus placebo (physiologic serum) before NGT insertion in patient needing enteral nutrition, using visual analogue scale. Secondary objectives are to evaluate nurse and patient satisfaction using questionnaires, facility of NGT insertion using Likert scale, numbers of try, time of procedure, complications like tracheal insertion and success of the insertion using thorax x-ray.

The study will be held in CHU Nice at nutrition unit support. After signed consentment, patients will be separate in two groups : group A (lidocaïne spray 5 %) and group B (physiologic serum). There will be 2 spray in nostril and 2 in orophagyngeal cavity 2 minutes before NGT insertion, which will be done by a competent nurse. Vital signs will be noted at the beginning of the procedure and 10 minutes after. At the end, the nurse and the patient will have to answer a questionnaire. Pain will be grade using visual analogue scale immediately after the procedure. Demographic data and complications will be note by the investigator. Finally, thorax X-ray will be done at the end of the procedure. There will be 34 patients by group. If the investigators find a benefit, this can change their practice and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Patient needing enteral nutrition by NGT
* Signed consentment
* Affiliation to securite sociale

Exclusion Criteria

* Lidocaine allergy
* Severe demencia
* Non cooperating patient
* Facial trauma and basal skull fracture
* Reflex deglutition problem
* Pulmonary illness like severe asthma
* Hemodynamic instability
* Pregnancy and nursing
* Patient on guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
EVA | one time
  Pain and comfort during NGT insertion will be evaluate using visual analogue scale (0 to 100 mm marqued at each side: extreme pain and no pain).

SECONDARY OUTCOMES:
Scales | one time
  * Nurse satisfaction using Likert scale from 1 to 5
  * Patient satisfaction using Likert scale from 1 to 5
  * Facility of NGT insertion using Likert scale from 1 to 5 and numbers of try: defined by numbers of insertions necessary by 1 operator.
  * Tolerance of the procedure: all complications will be note from beginning until 20 minutes.
  * Time for the NGT insertion defined like the number of minutes between the first attempt (when the nurse take the tube) until the end of the procedure.
  * Success of the insertion, defined by good insertion confirmed by an X-ray and procedure done by one operator.

CONTACTS AND LOCATIONS:
Overall Officials: GOMERCIC Cecile, Ph, Principal Investigator — CHU de Nice, Hôpital Archet, Pôle Digestif, 151 route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France